CLINICAL TRIAL: NCT05106400
Title: Open-label, Randomized, Four-treatment, Four-sequence, Four-period, Crossover, Single-application Study Evaluating and Comparing Product Adhesion in Healthy Adult Subjects Using ZTlido 1.8% Versus Salonpas(Lidocaine Patch 4%), Aspercreme(Lidocaine Patch 4%) and IcyHot(Lidocaine 4% + Menthol 1% Patch)
Brief Title: Clinical Adhesion Study Between ZTlido 1.8% and Three Over-the-counter External Analgesic Lidocaine-containing Patches
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A21.1463
Record Dates: First submitted 2021-10-11; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Healthy
MeSH Terms: interventions — Lidocaine; Capsaicin; trolamine salicylate; Menthol; Transdermal Patch

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to ZTlido (Lidocaine Topical System) 1.8% or Salonpas (Lidocaine Patch 4%) or Aspercreme (Lidocaine Patch 4%) or IcyHot (Lidocaine 4% + Menthol 1% Patch). Subjects will crossover to each treatment after a wash out period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ZTlido (Lidocaine Topical System) 1.8% (Other)
  Interventions: Drug: ZTlido (Lidocaine Topical System) 1.8%
- Salonpas (Lidocaine Patch 4%) (Other)
  Interventions: Drug: Salonpas (Lidocaine Patch 4%)
- Aspercreme (Lidocaine Patch 4%) (Other)
  Interventions: Drug: Aspercreme (Lidocaine Patch 4%)
- IcyHot (Lidocaine 4% + Menthol 1% Patch) (Other)
  Interventions: Drug: IcyHot (Lidocaine 4% + Menthol 1% Patch)

INTERVENTIONS:
Drug: ZTlido (Lidocaine Topical System) 1.8% — 1 ZTlido (Lidocaine Topical System) 1.8% is applied predetermined area on the right or left side of the mid to upper back and worn for 12 hours
  Arms: ZTlido (Lidocaine Topical System) 1.8%
Drug: Salonpas (Lidocaine Patch 4%) — 1 Salonpas (Lidocaine Patch 4%) is applied predetermined area on the right or left side of the mid to upper back and worn for 12 hours
  Arms: Salonpas (Lidocaine Patch 4%)
Drug: Aspercreme (Lidocaine Patch 4%) — 1 Aspercreme (Lidocaine Patch 4%) is applied predetermined area on the right or left side of the mid to upper back and worn for 12 hours
  Arms: Aspercreme (Lidocaine Patch 4%)
Drug: IcyHot (Lidocaine 4% + Menthol 1% Patch) — 1 IcyHot (Lidocaine 4% + Menthol 1% Patch) is applied predetermined area on the right or left side of the mid to upper back and worn for 12 hours
  Arms: IcyHot (Lidocaine 4% + Menthol 1% Patch)

SUMMARY:
The study is designed to evaluate and compare the clinical adhesion performance of the ZTlido (Lidocaine Topical System) 1.8% of Scilex Pharmaceuticals Inc. (Reference) versus Salonpas (Lidocaine Patch 4%), Aspercreme (Lidocaine Patch 4%) and IcyHot (Lidocaine 4% + Menthol 1% Patch), on the Mid to upper back while being worn for 12 hours in healthy adult human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male and female subjects aged 18 years and older with a Body Mass Index (BMI) range 18.0-32.49 kg/m2 inclusive (according to the formula of BMI = weight (kg) / [height (m)2]).
* Subjects who have no evidence of underlying disease during screening and check-in and whose screening is performed within 28 days of check-in.
* Subjects whose screening laboratory values are within normal limits or considered by the physician or Principal Investigator to be of no clinical significance.
* Absence of disease markers of HIV 1 & 2, hepatitis B & C virus.
* Generally healthy as documented by the medical history, physical examination (including but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory, musculoskeletal and central nervous systems) and vital sign assessments.
* Generally healthy as documented by 12-lead electrocardiogram (ECG), and clinical laboratory assessments.
* Any abnormalities/deviations from the acceptable range of medical history, clinical laboratory values, ECG and vitals, that might be considered clinically relevant by the study physician or investigator will be evaluated as individual cases.
* Subjects able to comply with study procedures, in the opinion of the Principal Investigator.
* Willing to give written consent and adhere to all the requirements of this protocol.
* Female subjects of childbearing potential;
* Non-pregnant and non-lactating females practicing medically acceptable forms of Birth Control and willing to continue during the study.
* Postmenopausal Female- Age > 45 years and Amenorrhea for at least 1 year; or Bilateral Oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months; or Total hysterectomy and an absence of bleeding for at least 3 months.
* Male volunteers must practice protected sex throughout the study.

Exclusion Criteria:

* Evidence of allergy or known hypersensitivity to lidocaine, local anesthetics of the amide type e.g., bupivacaine, etidocaine, mepivacaine and prilocaine or to any of the components of formulation.Any major illness in the last three months or any significant chronic medical illness.
* Subjects with history of addiction, abuse, and misuse of any drug - as per physician discretion.
* Subjects with history of mental illness as per physician discretion.
* Presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, hepatic, dermatologic, musculoskeletal, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease (as determined by the Medical Investigator).
* Participation in any clinical trial within 30 days prior to product application.
* Subjects with inflamed or injured skin, such as active herpes zoster lesions, atopic dermatitis or wounds where the product will be placed.
* Presence of any skin condition such as scratches, cuts, scars, abrasions, excessive hair, tattoos, moles, recently shaved skin, uneven skin texture, open sores, irritated (redness, rash, or blisters, etc.) or excessively oily skin at the application areas that may affect the application of the study product.
* Use of make-up, creams, lotions, powders, or other topical products to the skin area where the product will be placed, within 48 hours prior to product application.
* Use of antihistamines at product application site within 72 hours prior to product application.
* Using antiarrhythmic drugs (such as tocainide and mexiletine) and local anesthetics within 14 days prior to product application.
* Radiation therapy within 3 weeks prior to product application
* History of significant dermatologic cancers (e.g., melanoma, squamous cell carcinoma etc.) except basal cell carcinomas that were superficial and did not involve the investigative sites.
* Use of nicotine containing products (including e-cigarettes, patches, gum, chewing tobacco, cigars, etc.) within 30 days prior to patch application.
* Positive results for drugs of abuse and alcohol breath analysis prior to product application.
* Female subjects:
* Demonstrating a positive pregnancy screen
* Who are currently breastfeeding
* Use of hormone replacement therapy within three months prior to product application.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Change in Percent adhesion | 0, 3, 6, 8, 10, and 12 hours
  The adhesion performance (i.e., degree of lifting or detachment) is assessed by clinicians at each time point. The adhesion of Test Products 1, 2, and 3 (each over-the-counter external analgesic lidocaine-containing patch) are compared to the adhesion performance observed for the Reference Product.

SECONDARY OUTCOMES:
Adverse events | 12 hours
  The number of adverse events observed in each treatment will be used to assess the safety and tolerability of the four interventions

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Lissin, MD, Study Director — Chief Medical Officer
Locations (1):
- AXIS Clinicals, Dilworth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No